CLINICAL TRIAL: NCT06648707
Title: Dual-task Training to Prevent Cognitive Decline in Community-dwelling Older Adults: A Pilot Pragmatic Randomised Controlled Trial
Brief Title: Dual-task Training to Prevent Cognitive Decline in Community-dwelling Older Adults: A Pilot Pragmatic RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Health and Medical Research Fund (Other Government)
Responsible Party: Principal Investigator, Dr. Pui-Hing Chau, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UW 23-575
Record Dates: First submitted 2024-10-11; First posted 2024-10-18 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Community-dwelling Seniors
Keywords: dual-task; cognitive training; Older adults; train-the-trainer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Assigned intervention (Other): The intervention group will start 6 week dual-task invention immediately after baseline.
  Interventions: Other: Dual-task training
- Assigned waitlist control (Other): The control group will start 6 week dual-task invention after the follow-up assessment 6 weeks after baseline.
  Interventions: Other: Dual-task training

INTERVENTIONS:
Other: Dual-task training — Participants will receive a one-hour face-to-face group-based dual-task training session twice a week for 6 weeks. Training included cognitive components and physical components to be conducted simultaneously.

SUMMARY:
Objectives:

This study aims to explore the feasibility and acceptance of group-based dual-task training for prevention of cognitive decline in a pragmatic setting for community-dwelling older adults.

The primary objective is to assess recruitment rate, attendance rate, retention rate and satisfaction rate of participants.

Study design and participants:

This is a pilot pragmatic RCT with waitlist control. First, a co-design approach will be adopted to develop the intervention with the older adults. Then, about six participating community centres will nominate staff or volunteer to receive the training in order to lead the intervention. Informed consent will be sought from the participants and baseline assessment will be conducted. The participants will be randomly allocated to the intervention and control groups in 1:1 ratio using block randomisation with varying block size. At the end of the study, one representative of each participating centre will be invited to provide qualitative feedback.

Measurements:

The primary outcomes are the feasibility outcomes, namely the recruitment rate, attendance rate, the retention rate, and satisfaction rate of participants. Secondary outcomes include completion rate of the interventionist, time to recruit target sample size, factors influencing older adults' decision to participate and staff of the community centre to organise the activity, subjective memory complaints, working memory, executive function, and cognitive status of participants. A structured questionnaire will be used to collect quantitative outcomes related to effects and satisfaction. Qualitative feedback from representatives of the elderly community centres will be collected according to a semi-structured interview guide.

Expected results: The intervention is feasible and highly accepted by the participants and staff of the community centres. Potential effect-related outcomes are to be demonstrated.

ELIGIBILITY:
Inclusion Criteria:

(i) aged 65 years and above,

(ii) eligible to enrol in activities organised by the community centres,

(iii) no communication problems,

(iv) able to understand and follow instructions,

(v) able to read and write Chinese.

Exclusion Criteria:

contraindications to chair-based or stepping exercises.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | After baseline, before randomization
  Recruitment rate is defined as the number of participants agreed to join the study before randomization divided by the number of potential participants who completed recruitment briefing.
Attendance rate | 6 weeks after baseline for intervention group, 12 weeks after baseline for waitlist control group.
  Attendance rate is defined as the number of attended intervention sessions collected in attendance log divided by the number of planned intervention sessions.
Retention rate | 6 weeks after baseline for intervention group, 12 weeks after baseline for waitlist control group.
  Retention rate is defined as the number of participants completing the post-intervention assessment divided by the number of participants at baseline.
Satisfaction rate | 6 weeks after baseline for intervention group, 12 weeks after baseline for waitlist control group.
  Satisfaction to the project will be measured by a question using 5-point Likert scale (very satisfactory to very unsatisfactory). Satisfaction rate is defined as the number of participants rating the intervention a score of ≥4 out of 5 divided by the number of participants started intervention.

SECONDARY OUTCOMES:
Completion rate of the interventionist | End of study, up to 2 years
  The number of nominated staff/volunteers considered as completing the project divided by the total number of nominated staff/volunteers
Time to recruit target sample size | Before baseline
  The time needed to recruit target sample size is defined as the time taken to recruit required sample size in each centre.
Factors influencing older adults' decision to participate and staff of the community centre to organise the activity | At the end of recruitment briefing, before baseline
  Reasons of the older adults and staff of the community centres for joining or not joining the study
Change from baseline subjective memory complaints at 6 weeks | 6 weeks after baseline
  Subjective memory complaints will be measured by the 27-item Memory Inventory in Chinese (Lui et al., 2006). Participants response on the frequency of complaints related to daily living in the past month, using 0 (none) to 4 (continuously). The scale ranges from 0 to 108, higher score indicates more memory complaints.
Change from baseline subjective memory complaints at 12 weeks | 12 weeks after baseline, only for waitlist control group
  Subjective memory complaints will be measured by the 27-item Memory Inventory in Chinese (Lui et al., 2006). Participants response on the frequency of complaints related to daily living in the past month, using 0 (none) to 4 (continuously). The scale ranges from 0 to 108, higher score indicates more memory complaints.
Change from baseline working memory at 6 weeks | 6 weeks after baseline
  Working memory will be measured by Digit Span Test (Leung et al., 2011). The participants will repeat the digits series which are gradually longer. In both the forward and the backward test, the longer the series, the better the condition.
Change from baseline working memory at 12 weeks | 12 weeks after baseline, only for waitlist control group
  Working memory will be measured by Digit Span Test (Leung et al., 2011). The participants will repeat the digits series which are gradually longer. In both the forward and the backward test, the longer the series, the better the condition.
Change from baseline executive function at 6 weeks | 6 weeks after baseline
  Executive function will be measured by Chinese version of the Victoria Stroop Test (Lee and Chan, 2000). The completion time and number of errors that the participants made in naming the colour in the presence of different stimuli (number dots, words unrelated to color, words related to color) will be recorded, with more time and errors as worse condition.
Change from baseline executive function at 12 weeks | 12 weeks after baseline, only for waitlist control group
  Executive function will be measured by Chinese version of the Victoria Stroop Test (Lee and Chan, 2000). The completion time and number of errors that the participants made in naming the colour in the presence of different stimuli (number dots, words unrelated to color, words related to color) will be recorded, with more time and errors as worse condition.
Change from baseline cognitive status at 6 weeks | 6 weeks after baseline
  Cognitive status will be measured by the Montreal Cognitive Assessment 5-Minutes (Hong Kong Version) (HK-MoCA 5-Min) protocol. The validated assessment test covers four domains: attention, executive functions/language, orientation, and memory (Yeung et al., 2014). The total score ranges from 0 to 30; a higher score indicates better cognitive status.
Change from baseline cognitive status at 12 weeks | 12 weeks after baseline, only for waitlist control group
  Cognitive status will be measured by the Montreal Cognitive Assessment 5-Minutes (Hong Kong Version) (HK-MoCA 5-Min) protocol. The validated assessment test covers four domains: attention, executive functions/language, orientation, and memory (Yeung et al., 2014). The total score ranges from 0 to 30; a higher score indicates better cognitive status.
Qualitative feedback | At the end of the study, up to 2 years
  Qualitative feedback on facilitators and barriers of organising the activity will be collected from one representative of each participating centre by semi-structured interview.

CONTACTS AND LOCATIONS:
Overall Officials: Pui Hing Chau, PhD, Principal Investigator — School of Nursing, The University of Hong Kong
Locations (1):
- Community centre, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No